CLINICAL TRIAL: NCT05088863
Title: Survey Assessing How Consumers Adapt Their Diet in Response to Health Claim Messaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principal Investigator, St. Boniface Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS25165 (B2021:102); HS25165 (B2021:102) (Other: Biomedical research Ethics Board, University of Manitoba)
Record Dates: First submitted 2021-10-06; First posted 2021-10-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Health Claim Implementation
Keywords: health claim; flax
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implementation of health claim (Other): Participants will have 2 weeks to incorporate 40g of flaxseed per day into their diet
  Interventions: Other: flaxseed

INTERVENTIONS:
Other: flaxseed — 40g of flaxseed per day

SUMMARY:
A survey designed to examine how consumers adapt their diet in response to health claim messaging.

DETAILED DESCRIPTION:
384 participants will be recruited to participate (n=32/group) ensuring equal numbers based on gender (men and women), income (low and medium-high), and age (18-35, 36-55, >56 years). Participants will be asked to prepare a 3-day food record representative of their current dietary intake. Participants will then be told, "Health Canada has approved the following health claim: 40g of ground flaxseed per day has been shown to help lower cholesterol, which is a risk factor for heart disease." Without any further guidance, participants will then be asked to modify their diet to achieve 40g per day of flaxseeds for the following 2 weeks. They will be asked to prepare another 3-day food record so we can see if/how their diet changed. At the end of the 2-week period, participants will be asked if they were successful with the changes and what barriers they faced in implementing these changes. This survey will be accomplished remotely with informed consent and communication with participants happening over the phone or videoconference. Participants will mail the food records to clinical trial staff. Analysis of food records will identify the food choices used to achieve dietary change, if these changes altered nutrient intake compared to their usual diet and if they were able to achieve the target laid out (ie. 40g flaxseed per day). A questionnaire will be used to identify barriers to implementation of dietary change (ie. price, availability, sensory aspects of food, ease of preparation).

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman, age ≥18 years;
2. Willing to provide informed consent;
3. Willing/able to comply with the requirements of the study;
4. Have a mailing address in the Winnipeg census metropolitan area (City of Winnipeg and the municipalities of West St. Paul, East St. Paul, Headingley, Macdonald, Richot, Tache, Springfield, Rosser, St. Francois Xavier and St. Clements)4.

Exclusion Criteria:

1. Allergy, aversion or unwillingness to eat whole ground flaxseed;
2. Consuming ≥40g whole ground flaxseed/day;
3. A family member within the same household is participating or has participated in this study;
4. Currently participating in a food trial or dietary program that does not allow change in food choice.
5. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity fits into one of two categories, man or woman
Enrollment: 384 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
3-day food record to assess food choices to achieve health claim | Two weeks
  A list of flax containing foods from the 3-day food record will be created and the frequency with which each food item was selected will be recorded.
Comparison of 3-day food records to assess change in nutrient intake from usual diet to diet addressing health claim | Four weeks
  3 day food records before and after change in diet to address health claim will be entered into nutrition analysis software to calculate nutrient intake
Were they able to achieve the target laid out in the health claim | 2 weeks
  Questionnaire to identify barriers to implementation of health claim

SECONDARY OUTCOMES:
Barriers to implementation of dietary change | 2 weeks
  Questionnaire to identify if price, availability, sensory aspects of food, ease of preparation are barriers to implementation of the health claim

CONTACTS AND LOCATIONS:
Overall Officials: Heather Blewett, PhD, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- I. H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the time the data is collected until the manuscript is accepted for publication

REFERENCES:
- [Background] Kaur A, Scarborough P, Rayner M. A systematic review, and meta-analyses, of the impact of health-related claims on dietary choices. Int J Behav Nutr Phys Act. 2017 Jul 11;14(1):93. doi: 10.1186/s12966-017-0548-1. PMID 28697787
- See also: City of Winnipeg. Population of Winnipeg. April 2021: — https://www.winnipeg.ca/cao/pdfs/population.pdf
- See also: Statistics Canada. Table 11-10-0241-01 Low income cut-offs (LICOs) before and after tax by community size and family size, in current dollars DOI: — http://doi.org/10.25318/1110024101-eng
- See also: 5. Statistics Canada. Question #17 on the 2016 Census of Population 2A-L questionnaire: — https://www23.statcan.gc.ca/imdb/p3Instr.pl?Function=getInstrumentList&Item_Id=295122&UL=1V&
- See also: 2. Summary of Health Canada's Assessment of a Health Claim about Ground Whole Flaxseed and Blood Cholesterol Lowering — https://www.canada.ca/content/dam/hc-sc/migration/hc-sc/fn-an/alt_formats/pdf/label-etiquet/claims-reclam/assess-evalu/flaxseed-graines-de-lin-eng.pdf